CLINICAL TRIAL: NCT06390839
Title: MATCH Treatment Subprotocol Z1C: Phase II Study of Palbociclib (PD-0332991) in Patients With Tumors With CDK4 or CDK6 Amplification
Brief Title: Testing Palbociclib (PD-0332991) as Potentially Targeting Treatment in Cancers With CDK4 or CDK6 Amplification (MATCH - Subprotocol Z1C)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-01137; NCI-2024-01137 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-Z1C (Other: ECOG-ACRIN Cancer Research Group); EAY131-Z1C (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-04-27; First posted 2024-04-30 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm
MeSH Terms: conditions — Lymphoma | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (palbociclib) (Experimental): Patients receive palbociclib PO QD on days 1-21 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT or MRI and blood sample collection throughout the trial. Patients may also undergo a biopsy on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Palbociclib

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Palbociclib — Given PO
  Other Names: 6-Acetyl-8-cyclopentyl-5-methyl-2-((5-(piperazin-1-yl)pyridin-2-yl)amino)-8h-pyrido(2,3-d)pyrimidin-7-one; Ibrance; PD 0332991; PD 332991; PD 991; PD-0332991; PD0332991

SUMMARY:
This phase II MATCH treatment trial tests how well palbociclib (PD-0332991) works in treating patients with cancer that has certain genetic changes. Palbociclib (PD-0332991) is in a class of medications called kinase inhibitors. It is used in patients whose cancer has a certain mutation (change) in the CDK4 or CDK6 gene. It works by blocking the action of mutated CDK4 or CDK6 that signals cancer cells to multiply. This helps to stop or slow the spread of cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive palbociclib orally (PO) once daily (QD) on days 1-21 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo computed tomography (CT) or magnetic resonance imaging (MRI) and blood sample collection throughout the trial. Patients may also undergo a biopsy on study.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 1 year.

THE MATCH SCREENING TRIAL:

Please see NCT02465060 for information on the MATCH Screening Protocol and applicable documents.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol EAY131/ NCI-2015-00054 prior to registration to treatment subprotocol
* Patients must have CDK4 amplification or CDK6 amplification, or another aberration, as determined via the MATCH Master Protocol
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
* Patients must not have breast cancer, mantle cell lymphoma, myeloma, or liposarcoma
* Patients must not have known hypersensitivity to palbociclib or compounds of similar chemical or biologic composition
* Patients with known or symptoms of left ventricular dysfunction will be excluded
* Patients must not have received prior therapy with a CDK4 or CDK6 inhibitor (including but not limited to palbociclib, abemaciclib, or ribociclib)
* Patients must not be using drugs or foods that are known potent CYP3A4 inhibitors or inducers, or are CYP3A substrates with narrow therapeutic indices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mark H O'Hara, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol Z1C was activated on March 13, 2017. Forty-three patients were enrolled on EAY131-Z1C between March 2017 and June 2021. These patients were enrolled into 2 cohorts, a primary and an expansion cohort. The primary cohort enrolled 35 patients. This subprotocol was suspended in Oct, 2018 after meeting its original accrual goal of 35 patients. This subprotocol was reactivated in May, 2020 and subsequently closed on May 25, 2021, with 8 patients enrolled to the expansion cohort.
Pre-assignment Details: Out of the 43 patients, 16 patients were enrolled on the basis of the results from the NCI-MATCH assay and 27 on the basis of the outside assay results. Twelve of the 27 outside lab patients had their samples centrally confirmed.
Groups:
- Treatment (Palbociclib): Patients receive palbociclib 125mg PO QD on days 1-21 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT or MRI and blood sample collection throughout the trial. Patients may also undergo a biopsy on study.
Period: Overall Study
Arm/Group | Treatment (Palbociclib)
Started | 43
Started Protocol Therapy | 40
Eligible and Treated | 38
Eligible, Treated and Mutation Status Confirmed (Primary efficacy analysis set) | 25
Completed | 0
Not Completed | 43
Not completed — Ineligible | 2
Not completed — Never start protocol therapy | 3
Not completed — Adverse Event | 1
Not completed — Alternative therapy | 2
Not completed — Death | 3
Not completed — Disease progression | 28
Not completed — Withdrawal by Subject | 2
Not completed — Complicating disease | 1
Not completed — Noncompliance | 1

BASELINE CHARACTERISTICS:
Population: Patients who were eligible, started protocol therapy, and had mutation status confirmed at the analysis time were the analyzable patients
Arm/Group | Treatment (Palbociclib)
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 61 [25 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among analyzable patients. Objective response is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Details about how to define complete response and partial response can be found in the master protocol. 90% two-sided binomial exact confidence interval is calculated for ORR.
Time Frame: Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible, treated and mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Palbociclib)
Number analyzed (Participants) | 25
percentage of participants | 4 [0.2 to 17.6]

2. Secondary Outcome: 6-month Progression Free Survival (PFS) Rate
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until disease progression, up to 3 years post registration, from which 6-month PFS rate is determined
Population: Eligible, treated and mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Palbociclib)
Number analyzed (Participants) | 25
percentage of participants | 16.7 [7.9 to 35.3]

3. Secondary Outcome: Progression Free Survival
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible, treated and mutation status confirmed
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Palbociclib)
Number analyzed (Participants) | 25
months | 2 [1.8 to 2.2]

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years post registration.
Description: All patients enrolled were included in the all-cause mortality analysis. Forty patients were included in the toxicity analysis (excluding three who did not receive treatment).
Arm/Group | Treatment (Palbociclib)
All-Cause Mortality (participants affected / at risk) | 33/43
Serious Adverse Events (participants affected / at risk) | 22/40
Other Adverse Events (participants affected / at risk) | 30/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Palbociclib) (N=40)
Anemia (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Alkaline phosphatase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 8
Neutrophil count decreased (Investigations) | 14
Platelet count decreased (Investigations) | 2
White blood cell decreased (Investigations) | 10
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Palbociclib) (N=40)
Anemia (Blood and lymphatic system disorders) | 9
Fatigue (General disorders) | 17
Abdominal pain (Gastrointestinal disorders) | 2
Bloating (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 3
Alanine aminotransferase increased (Investigations) | 4
Alkaline phosphatase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 3
Creatinine increased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 17
Platelet count decreased (Investigations) | 13
White blood cell decreased (Investigations) | 17
Anorexia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Insomnia (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/39/NCT06390839/Prot_000.pdf